CLINICAL TRIAL: NCT01561144
Title: UMBRELLA - Incidence of Arrhythmias in Spanish Population With a Medtronic ICD Implant
Brief Title: UMBRELLA - Incidence of Arrhythmias in Spanish Population With a Medtronic Implantable Cardiac Defibrillator (ICD) Implant
Acronym: UMBRELLA
Status: Terminated | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: UMBRELLA
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cardiomyopathies; Cardiac Arrhythmias; Cardiac Arrest
Keywords: Defibrillators, Implantable; Cardiac arrhythmias; Heart Disease
MeSH Terms: conditions — Cardiomyopathies; Arrhythmias, Cardiac; Heart Arrest; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
The purpose of the study is to analyze the different patient profiles implanted with an Implantable Cardiac Defibrillator (ICD) in Spain (guidelines adoption) and the patient prognosis as a function of clinical profile, implant indication, arrhythmias incidence, treatments or device programming.

DETAILED DESCRIPTION:
Umbrella is a prospective and retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Medtronic Implantable Cardiac Defibrillator (ICD) according to guidelines.
* Patients with CareLink home Telemonitoring System.

Exclusion Criteria:

* Unwillingness or inability to sign study written informed consent and/or CareLink consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients inplanted with an Implantable Cardiac Defibrillator (ICD) according to guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 4648 (Actual)
Dates: Start 2011-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
To assess the number of ventricular and atrial arrhythmias, and atrial fibrillation burden detected by ICD. | End of the study, an expected duration of 5 years.

CONTACTS AND LOCATIONS:
Locations (51):
- Spain (51):
  - H. General Universitario de Elche, Elche, Alicante
  - H. de Txagorritxu, Vitoria-Gasteiz, Araba
  - H. Universitari Germans Trias i Pujol, Badalona, Barcelona
  - H. Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario de Santiago, Santiago de Compostela, Coruña
  - Complejo Hospitalario Donostia, Donostia / San Sebastian, Guipúzcoa
  - H. Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - H. Rafael Méndez, Lorca, Murcia
  - H. Universitario Central de Asturias, Oviedo, Principality of Asturias
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - H. Universitario De La Ribera, Alzira, Valencia
  - H. de Cruces, Barakaldo, Vizcaya
  - H. Galdakao - Usansolo, Galdakao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - H. General de Alicante, Alicante
  - H. Universitario San Juan de Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas de Almería, Almería
  - H. Infanta Cristina, Badajoz
  - H. Clinic I Provincial de Barcelona, Barcelona
  - H. de la Santa Creu i Sant Pau, Barcelona
  - H. de Basurto, Bilbao
  - H. Universitario de Burgos, Burgos
  - Complejo Hospitalario de Cáceres, Cáceres
  - H. San Pedro de Alcántara, Cáceres
  - H. Gral de Ciudad Real, Ciudad Real
  - H. Reina Sofía, Córdoba
  - H.Universitario Virgen de las Nieves, Granada
  - H.Universitario de Guadalajara, Guadalajara
  - H. Universitario Insular de las Palmas, Las Palmas de Gran Canaria
  - H. De León, León
  - H. Clínico San Carlos, Madrid
  - H. Infanta Leonor, Madrid
  - H. Universitario 12 de Octubre, Madrid
  - H. Universitario Gregorio Marañón, Madrid
  - H. Universitario La Paz, Madrid
  - H. Universitario Ramón y Cajal, Madrid
  - H. Clínico Virgen de la Victoria, Málaga
  - H. General Universitario Reina Sofía, Murcia
  - H. Universitario Virgen de la Arrixaca, Murcia
  - H. Son Llátzer, Palma de Mallorca
  - H. de Navarra, Pamplona
  - H.Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - H. Universitario Marqués de Valdecilla, Santander
  - H. Universitario Nuestra Señora de Valme, Seville
  - H. Universitario Virgen Macarena, Seville
  - H. Universitario Joan XXIII, Tarragona
  - Complejo Hospitalario de Toledo, Toledo
  - H. General Universitario de Valencia, Valencia
  - H. Universitario la Fe, Valencia
  - H. Clínico Universitario de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo

REFERENCES:
- [Derived] Briongos-Figuero S, Garcia-Alberola A, Rubio J, Segura JM, Rodriguez A, Peinado R, Alzueta J, Martinez-Ferrer JB, Vinolas X, Fernandez de la Concha J, Anguera I, Martin M, Cerda L, Perez L; UMBRELLA Investigators *. Long-Term Outcomes Among a Nationwide Cohort of Patients Using an Implantable Cardioverter-Defibrillator: UMBRELLA Study Final Results. J Am Heart Assoc. 2021 Jan 5;10(1):e018108. doi: 10.1161/JAHA.120.018108. Epub 2020 Dec 25. PMID 33356406
- [Derived] Loughlin G, Datino T, Arenal A, Ruiz-Granell R, Sanchez-Gomez JM, Perez L, Martinez-Ferrer J, Alzueta J, Perez-Lorente F, Vinolas X, Fidalgo Andres ML, Fernandez de la Concha J. Predictors of adoption and impact of evidence-based programming on the incidence of implantable cardioverter-defibrillator therapies. Rev Esp Cardiol (Engl Ed). 2021 Apr;74(4):296-302. doi: 10.1016/j.rec.2020.06.017. Epub 2020 Aug 6. English, Spanish. PMID 32773348
- [Derived] Lillo-Castellano JM, Marina-Breysse M, Gomez-Gallanti A, Martinez-Ferrer JB, Alzueta J, Perez-Alvarez L, Alberola A, Fernandez-Lozano I, Rodriguez A, Porro R, Anguera I, Fontenla A, Gonzalez-Ferrer JJ, Canadas-Godoy V, Perez-Castellano N, Garofalo D, Salvador-Montanes O, Calvo CJ, Quintanilla JG, Peinado R, Mora-Jimenez I, Perez-Villacastin J, Rojo-Alvarez JL, Filgueiras-Rama D. Safety threshold of R-wave amplitudes in patients with implantable cardioverter defibrillator. Heart. 2016 Oct 15;102(20):1662-70. doi: 10.1136/heartjnl-2016-309295. Epub 2016 Jun 13. PMID 27296239
- [Derived] Anguera I, Dallaglio P, Martinez-Ferrer J, Rodriguez A, Alzueta J, Perez-Villacastin J, Porres JM, Vinolas X, Fontenla A, Fernandez-Lozano I, Garcia-Alberola A, Sabate X. Shock Reduction With Multiple Bursts of Antitachycardia Pacing Therapies to Treat Fast Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter Defibrillators: A Multicenter Study. J Cardiovasc Electrophysiol. 2015 Jul;26(7):774-82. doi: 10.1111/jce.12699. Epub 2015 May 28. PMID 25916814